CLINICAL TRIAL: NCT05862220
Title: A Single-center Study for the Correlation Between Computer Tomography Angiography and D-Dimer Level for the Diagnosis of Pulmonary Embolism
Brief Title: Correlation Between Computer Tomography Angiography and D-Dimer Level for the Diagnosis of Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Zulekha Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: ZH-12-2022-01
Record Dates: First submitted 2023-04-26; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: D-Dimer as an Early Detector of Pulmonary Embolism
Keywords: D-Dimer, Pulmonary, Embolism, CTPA.
MeSH Terms: conditions — Embolism; Cataract, posterior polar, 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- D-Dimer group: A blood sample was taken before starting the patients on any thrombolytic treatment. The latex agglutination test was used to measure plasma D-dimer level; this was done using a Sysmex CA-7000 automatic coagulation unit. The positivity threshold was above 250 ng/ml.
  Interventions: Diagnostic Test: D-Dimer vs CTPA
- CTPA group: CTPA was performed after performing blood sampling using Siemens Somatom definition AS 24 slice scanners. Non-ionic water-soluble contrast Omnipaque 350 mg I/mg or Visipaque 320 mg I/mg was injected at 4 mm/s maximum dose 100 ml using a Medtron pressure injector.
  Interventions: Diagnostic Test: D-Dimer vs CTPA

INTERVENTIONS:
Diagnostic Test: D-Dimer vs CTPA — CTPA was performed after performing blood sampling using Siemens Somatom definition AS 24 slice scanners. Non-ionic water-soluble contrast Omnipaque 350 mg I/mg or Visipaque 320 mg I/mg was injected at 4 mm/s maximum dose 100 ml using a Medtron pressure injector.OR, A blood sample was taken before starting the patients on any thrombolytic treatment. The latex agglutination test was used to measure plasma D-dimer level; this was done using a Sysmex CA-7000 automatic coagulation unit. The positivity threshold was above 250 ng/ml.

SUMMARY:
A blood sample was taken before starting the patients on any thrombolytic treatment. The positivity threshold for D-Dimer was above 250 ng/ml. CTPA was performed after performing blood sampling. Patients with confirmed pulmonary embolisms were admitted to ICU for continued monitoring of vitals, consciousness level, and signs of tissue perfusion. Signs of shock or hemodynamic instability should be observed regularly. Patients were managed in the ICU with anticoagulants by parenteral use. The most commonly used items were Heparin, either Unfractionated (UFH) or low-molecular-weight heparin (LMWH).D-dimer levels can leverage to detect PE. D-dimer levels can help in guiding the option of CTPA and the initiation of treatment for patients with suspected PE.

DETAILED DESCRIPTION:
A blood sample was taken before starting the patients on any thrombolytic treatment. The positivity threshold for D-Dimer was above 250 ng/ml. CTPA was performed after performing blood sampling. Patients with confirmed pulmonary embolisms were admitted to ICU for continued monitoring of vitals, consciousness level, and signs of tissue perfusion. Signs of shock or hemodynamic instability should be observed regularly. Patients were managed in the ICU with anticoagulants by parenteral use. The most commonly used items were Heparin, either Unfractionated (UFH) or low-molecular-weight heparin (LMWH).Presenting symptoms were mainly dyspnea, chest pain or discomfort, cough, and shortness of breath. Twenty-four patients of the total number of cases were positive for CTPA while four patients were negative for PE by CTPA. embolism was detected in the anterior, posterior, medial, and lateral basal segmental branches of the right lung, the lateral, posterior, and anterior basal segmental branches of the left lung, and the posterior segmental branch of the left lung. The D-dimer test and CTPA both provided similarly accurate PE diagnoses with no significant differences between them. There were 28 patients total, 3 of those patients had D-dimer levels below the cut-off value of 250 ng/ml, whereas the remaining 25 had D-dimer levels over the diagnostic threshold. Those with a positive CTPA diagnosis of PE had greater levels of D dimers than those with a negative CTPA diagnosis of PE. plasma D-dimer concentration did not correlate with the cross-sectional diameter of the blocked pulmonary vessel.D-dimer levels can leverage to detect PE. D-dimer levels can help in guiding the option of CTPA and the initiation of treatment for patients with suspected PE.

ELIGIBILITY:
Inclusion Criteria: Acute chest pain, dyspnea, tachypnea, and suspicion of PE -

Exclusion Criteria:the history of PE, the administration of anticoagulant medication before blood sampling, an allergic response to the CTPA contrast agent, impaired hepatic function or renal function, inability to cooperate during examinations, and an absence of relevant medical records for analyses

-

Ages: 22 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 28 patients included, 14 patients female and 14 patients of male gender with an average age of 55.4 ±11.2 years. Presenting symptoms were mainly dyspnea, chest pain or, cough, and shortness of breath. Twenty-four patients of the total number of cases were positive for CTPA while four patients were negative for PE by CTPA. No allergy to the contrast was recorded during our study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
the robustness of d-dimer testing for PE compared to CTPA and identify the threshold values to support its use | 26 MONTHS
  the study aims to ascertain the robustness of d-dimer testing for PE compared to CTPA and identify the threshold values to support its use

CONTACTS AND LOCATIONS:
Overall Officials: helena elizabith, consultant, Study Chair — Zulekha Hospitals
Locations (1):
- Zulekha Hospitals, Dubai, United Arab Emirates